CLINICAL TRIAL: NCT00042250
Title: Cell Cycle Kinetics in Vivo in Patients With Hematologic Malignancies Studied by Iododeoxyuridine and Bromodeoxyuridine Labelling
Brief Title: IUdR/BUdR Cell Cycle Labelling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DM91-102
Record Dates: First submitted 2002-07-24; First posted 2002-07-26 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Hematologic Malignancies
Keywords: Cell Cycle Interphase; G0; G1; G2; S Phase
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Chemotherapy for hematologic malignancy

SUMMARY:
To determine cell cycle parameters and changes after treatment, the labelling agent is given and a bone marrow aspiration is accomplished before treatment and after treatment for comparison. Participants must be undergoing concurrent therapy for hematologic malignancy.

DETAILED DESCRIPTION:
Cell cycle parameters include LI, Ts, Tc, T dpot, changes in these parameters, and differences between normal and leukemic cells in patients with hematologic malignancy prior to and following treatment.

ELIGIBILITY:
Histologic proof of one of:

* AML, ALL, or AUL
* MDS or CMML
* CML
* OR undergoing bone marrow transplantation.

Participants should be:

* off therapy for at least two weeks
* At least 18 years old or older
* Using adequate contraception if of child-bearing capability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 1992-05; Primary Completion 2002-10 (Actual); Study Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Andreeff, MD, PhD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M. D. Anderson Cancer Center — http://www.mdanderson.org